CLINICAL TRIAL: NCT00455013
Title: A Randomized, Open-Label, Multicenter, Parallel-Group Study of Belatacept (BMS-224818)-Based Corticosteroid-Free Regimens in Renal Transplant
Brief Title: A Phase II Study of Belatacept (BMS-224818) With a Steroid-free Regimen in Subjects Undergoing Kidney Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM103-034
Record Dates: First submitted 2007-03-30; First posted 2007-04-02 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: Kidney transplant
MeSH Terms: interventions — thymoglobulin; Abatacept; Sirolimus; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- belatacept, mycophenolate mofetil (MMF) (Experimental): thymoglobulin 1.5mg/kg for 4 days;IV belatacept: 10 mg/kg Days 1 and 5, then every other week through Month 3 (Weeks 2,4,6,8,10,12), and then every 4 weeks through Month 6 (Weeks 16, 20, 24),after 6 months, 5 mg/kg every 4 weeks until 12 months; MMF 1g twice daily(bis in die, BID)
  Interventions: Drug: Thymoglobulin; Drug: Belatacept; Drug: Mycophenolate Mofetil (MMF)
- belatacept, sirolimus (Experimental): thymoglobulin 1.5mg/kg for 4 days;IV belatacept: 10 mg/kg Days 1 and 5, then every other week through Month 3 (Weeks 2,4,6,8,10,12), and then every 4 weeks through Month 6 (Weeks 16, 20, 24),after 6 months, 5 mg/kg every 4 weeks until 12 months;sirolimus 5 mg/day on Day 1 (day of transplant)and continued through Day 2, dosing to be adjusted to keep pre-dose C0 levels at 7-12 ng/mL for first 6 months, followed by 5 - 10 ng/mL until 12 months.
  Interventions: Drug: Thymoglobulin; Drug: Belatacept; Drug: Sirolimus
- tacrolimus, MMF (Other): (IMPs as comparator regimen)thymoglobulin 1.5mg/kg for 4 days; oral tacrolimus 0.1 mg/kg/day in 2 divided doses with initial targeted trough level of 8-12 ng/mL for Days 1 - 30 with dose reduction to achieve 12 hour trough target of 5-10 ng/mL for 12 months; MMF (mycophenolate mofetil) 1g BID.
  Interventions: Drug: Thymoglobulin; Drug: Tacrolimus; Drug: Mycophenolate Mofetil (MMF)

INTERVENTIONS:
Drug: Thymoglobulin — Induction therapy, IV infusion, All subjects will receive thymoglobulin 1.5-mg/kg i.v. infusion on Days 1 (day of transplant), 2, 3, and 4 (up to a maximum total dose of 6 mg/kg) i.v. infusion over at least 4 hours
Drug: Belatacept — Belatacept arms will receive i.v. belatacept (10 mg/kg) on Days 1 and 5, and then every other week through Month 3 (Weeks 2, 4, 6, 8, 10, and 12), and then every 4 weeks through Month 6 (Weeks 16, 20, and 24). After 6 months, subjects will receive belatacept at the maintenance dose of 5 mg/kg every 4 weeks until completion of the trial
  Other Names: BMS-224818
  Arms: belatacept, mycophenolate mofetil (MMF); belatacept, sirolimus
Drug: Sirolimus — Sirolimus will be initiated at 5 mg/day on Day 1 (day of transplant) and continued through Day 2. The dosing will be adjusted subsequently to keep pre-dose (C0) levels at 7 - 12 ng/mL for the first 6 months, followed by 5 - 10 ng/mL thereafter
  Arms: belatacept, sirolimus
Drug: Tacrolimus — The recommended total initial dose of tacrolimus is 0.1 mg/kg/day in two divided doses orally up to and including week 52. Post week 52 subjects assigned to the tacrolimus arm will receive tacrolimus orally in accordance with local practice and the package insert until completion of the trial
  Arms: tacrolimus, MMF
Drug: Mycophenolate Mofetil (MMF) — Administered orally in a capsule or solution formulation in 2 divided doses on a consistent schedule in relation to time of day and meals. The dose should be 1 g bid; however 1.5 g bid may be administered at the investigator's discretion until completion of the trial
  Arms: belatacept, mycophenolate mofetil (MMF); tacrolimus, MMF

SUMMARY:
The purpose of this clinical research study is to learn if belatacept (BMS-224818) is expected to show acceptable rates of acute rejection (AR) in steroid-free belatacept-based immunosuppressive regiments compared to a similar steroid-free tacrolimus regimen. The long-term safety and tolerability of belatacept based regimens following long-term administration in subjects who have received a kidney transplant

ELIGIBILITY:
Inclusion Criteria:

* Living or deceased donor renal allograft
* Men and women, 18 to 70 years old
* Subjects who have received a de novo kidney transplant, who have completed the initial study treatment through Month 12, and are willing to sign informed consent will be eligible to continue into the long term extension phase

Exclusion Criteria:

* Pregnant or breastfeeding women
* Epstein Barr Virus (EBV) negative serology
* First time renal transplant with panel reactive antibody (PRA) ≥ 50% or retransplantation with PRA > 30%
* Graft loss due to AR
* Positive T-cell or B-cell crossmatch
* Recipients/donors with HIV or hepatitis B/C
* Active tuberculosis (TB)
* Immunosuppressive therapy within 1 year of enrollment
* UNOS ECD organs will be excluded
* Body mass index (BMI) > 35 kg/m²
* Subjects who have developed any malignancy (other than non-melanoma skin cancer) or other medical condition that, in the investigator's opinion, should not be treated with an experimental immunosuppressive drug like belatacept

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (11):
  - Ucsf, San Francisco, California
  - Denver Nephrology, Pc, Denver, Colorado
  - University Of Colorado Health Sciences Center, Denver, Colorado
  - Medical College Of Georgia, Augusta, Georgia
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - Henry Ford Hospital, Detriot, Michigan
  - Albany Medical College, Albany, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - University Of Cincinnati, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Italy (4):
  - Local Institution, Bologna, Bologna
  - Local Institution, Brescia
  - Local Institution, Padua
  - Local Institution, Roma
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Seville

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First 6 months (July 2007 to October 2008) assessed acute rejection of the renal transplant up to that time. All outcome measures were also assessed at 12 months post transplantation. Participants who wished to continue into the long term extension (LTE) signed a new consent form and were evaluated at 24, 36, and 48 Months post transplantation.
Pre-assignment Details: Epstein-Barr virus positive recipients of renal allograft from living or deceased donor. Excluded if panel reactive antibodies greater than, equal to (>=) 50 % or prior graft loss due to acute rejection. 93 participants randomized; 89 transplanted/treated: (1) fever on the day of surgery, (1) problem with allograft, and (2) withdrawal of consent.
Groups:
- Belatacept, Mycophenolate Mofetil (MMF): Thymoglobulin 1.5mg/kg for 4 days plus 4 corresponding doses of corticosteroids; intravenous infusion (IV) belatacept: 10 milligram per kilogram of weight (mg/kg) Day 1 (day of transplant) and Day 5, then every other week through Month 3 (Weeks 2,4,6,8,10,12), and then every 4 weeks through Month 6 (Weeks 16, 20, 24), after 6 months, 5 mg/kg every 4 weeks until 12 months; MMF (mycophenolate mofetil) 1g twice daily(BID). Participants were allowed to switch from MMF to sirolimus. Background immunosuppressive medications: methylprednisolone administered as 500, 250, 125, and 60 mg IV on Days 1, 2, 3, 4; thymoglobulin 1.5 mg/kg IV infusion on Days 1 (day of transplant), 2, 3, 4, up to maximum dose of 6 mg/kg.
- Belatacept, Sirolimus: Thymoglobulin 1.5mg/kg for 4 days plus 4 corresponding doses of corticosteroids; IV belatacept: 10 mg/kg Days 1 and 5, then every other week through Month 3 (Weeks 2, 4, 6, 8, 10, 12), and then every 4 weeks through Month 6 (Weeks 16, 20, 24),after 6 months, 5 mg/kg every 4 weeks until Month 12; sirolimus 5 mg/day on Day 1 and continued through Day 2, dosing to be adjusted to keep pre-dose C0 (concentration at time zero after administration) levels at 7-12 nanograms per milliliter (ng/mL) for first 6 months, followed by 5 - 10 ng/mL until 12 months. Participants were allowed to switch from sirolimus to MMF. Background immunosuppressive medications: methylprednisolone was administered as 500, 250, 125, and 60 mg IV on Days 1, 2, 3, 4, up to maximum dose of 6 mg/kg.
- Tacrolimus, MMF: Comparator regimen: thymoglobulin 1.5mg/kg for 4 days plus 4 corresponding doses of corticosteroids; oral tacrolimus 0.1 mg/kg/day in 2 divided doses with initial targeted trough level of 8-12 ng/mL for Days 1 - 30 with dose reduction to achieve 12 hour trough target of 5-10 ng/mL for 12 months; MMF 1g BID. Background immunosuppressive medications: methylprednisolone administered as 500, 250, 125, and 60 mg IV on Days 1, 2, 3, 4; thymoglobulin 1.5 mg/kg IV infusion on Days 1, 2, 3, 4 up to maximum dose of 6 mg/kg.
Period: Short Term Period
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Started | 33 (35 randomized, 33 transplanted and treated.) | 26 (27 randomized, 26 transplanted and treated.) | 30 (31 randomized, 30 transplanted and treated)
Completed | 27 (5 discontinued belatacept by Month 6 (1 more by Month 12), 2 switched from MMF to sirolimus.) | 21 (5 discontinued belatacept by Month 6; 10 additional switched from sirolimus to MMF.) | 28 (1 discontinued tacrolimus by Month 6 and 2 discontinued by Month 12 (1 more by Month 12))
Not Completed | 6 | 5 | 2
Not completed — Adverse Event | 2 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lack of Efficacy | 4 | 0 | 0
Not completed — Other | 0 | 0 | 1
Period: Long Term Extension (LTE)
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Started | 27 | 19 (2 Participants chose not to enter the LTE.) | 27 (1 Participant chose not to enter the LTE.)
Completed | 25 | 16 | 20
Not Completed | 2 | 3 | 7
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Death | 1 | 1 | 0
Not completed — No longer met criteria | 0 | 0 | 1
Not completed — Subject Request or refused | 0 | 0 | 3
Not completed — Poor non-compliance | 0 | 1 | 0
Not completed — non-specified | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received transplant and were treated with drug were analyzed up to Month 12 post transplant.
Groups:
- Belatacept, Mycophenolate Mofetil (MMF): Thymoglobulin 1.5mg/kg for 4 days plus 4 corresponding doses of corticosteroids; IV belatacept: 10 mg/kg Days 1 and 5, then every other week through Month 3 (Weeks 2, 4, 6, 8, 10, 12), and then every 4 weeks through Month 6 (Weeks 16, 20, 24), after 6 months, 5 mg/kg every 4 weeks until Month 12; MMF 1g BID. Participants were allowed to switch from MMF to sirolimus.
- Belatacept, Sirolimus: Thymoglobulin 1.5mg/kg for 4 days plus 4 corresponding doses of corticosteroids; IV belatacept: 10 mg/kg Days 1 and 5, then every other week through Month 3 (Weeks 2, 4, 6, 8, 10, 12), and then every 4 weeks through Month 6 (Weeks 16, 20, 24),after 6 months, 5 mg/kg every 4 weeks until Month 12; sirolimus 5 mg/day on Day 1 and continued through Day 2, dosing to be adjusted to keep pre-dose C0 (concentration at time zero after administration) levels at 7-12 ng/mL for first 6 months, followed by 5 - 10 ng/mL until Month 12. Participants were allowed to switch from sirolimus to MMF.
- Tacrolimus, MMF: Comparator regimen: thymoglobulin 1.5mg/kg for 4 days plus 4 corresponding doses of corticosteroids; oral tacrolimus 0.1 mg/kg/day in 2 divided doses with initial targeted trough level of 8-12 ng/mL for Days 1 - 30 with dose reduction to achieve 12 hour trough target of 5-10 ng/mL for 12 months; MMF (mycophenolate mofetil) 1g BID.
- Total: Total of all reporting groups
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF | Total
Number analyzed (Participants) | 33 | 26 | 30 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 24 | 26 | 83
  >=65 years | 0 | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (11.1) | 52.7 (10.8) | 53.6 (13.2) | 51.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 8 | 22
  Male | 25 | 20 | 22 | 67
Region of Enrollment [Number; unit: participants]
  North America | 22 | 16 | 20 | 58
  Europe | 11 | 10 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Rejection (AR) of Transplant up to 6 Months Post Transplantation - Intent to Treat (ITT) Population
Description: AR is clinicopathological event requiring clinical evidence and biopsy confirmation by central pathologist. One or more conditions were met and a renal biopsy revealed histologic evidence of rejection: unexplained rise of serum creatine (SCr) greater than or equal to 25% from baseline plus one or more of the following: unexplained decreased urine output; fever, graft tenderness; SCr that remained elevated 14 days post-transplantation and clinical suspicion of AR; other reason and participant treated for episode. Day 1=transplantation. Banff 97 working classification of kidney transplant pathology: Type I=tubulointerstitial AR without arteritis (IA: interstitial infiltration with >25% of parenchyma affected and moderate tubulitis with >4 mononuclear cells/tubular cross section; IB: >10 mononuclear cells; Type II vascular AR with (IA) intimal arteritis (IIA=mild - moderate; IIB=severe; Type III=severe rejection with transmural arterial changes, necrosis of smooth muscle cells.
Time Frame: Day 1 to Month 6 post-transplantation
Population: Participants with more than one episode of AR were counted once only and the episode with the worst grade was used. For 95% Confidence Interval (CI) within each group, normal approximation was used if N greater than, or equal to (>=) 5. Otherwise, exact method was used. ITT population defined as all randomized and transplanted participants.
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 33 | 26 | 30
participants
  Total Number of Participants with AR | 4 [3.4 to 28.2] | 1 [0.1 to 19.6] | 1 [0.1 to 17.2]
  Mild Acute IA | 0 | 0 | 0
  Mild Acute IB | 0 | 0 | 0
  Moderate Acute IIA | 2 | 0 | 1
  Moderate Acute IIB | 1 | 1 | 0

2. Secondary Outcome: Number of Participants With Acute Rejection of Transplant up to Month 12 Post Transplantation - Intent to Treat Population
Description: AR defined as a clinicopathological event requiring clinical evidence and biopsy confirmation by central pathologist. One or more conditions were met and a renal biopsy revealed histologic evidence of rejection: unexplained rise of serum creatine (SCr) >= 25 % from baseline plus one or more of the following: unexplained decreased urine output; fever and graft tenderness; a SCr that remained elevated within 14 days after transplantation and clinical suspicion of AR; reason other than those listed and participant was treated for this episode. Day 1 was day of transplantation. Banff grade used Banff 97 working classification of kidney transplant pathology. ITT population was all randomized and transplanted participants.
Time Frame: Day 1 to Month 12 post transplantation
Population: For 95% CI within each group, normal approximation was used if N greater than, equal to 5. Otherwise, exact method was used.
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 33 | 26 | 30
participants
  Total number of participants with AR | 5 [2.9 to 27.4] | 1 [0.1 to 19.6] | 1 [0.1 to 17.2]
  Mild Acute IA | 0 | 0 | 0
  Mild Acute IB | 0 | 0 | 0
  Moderate Acute IIA | 3 | 0 | 1
  Moderate Acute IIB | 2 | 1 | 0

3. Secondary Outcome: Number of Participants With Graft Loss or Death up to Month 6 and Month 12 Post Transplantation - Intent to Treat Population
Description: Graft loss was defined as either functional loss or physical loss. Functional loss was defined as either: sustained level of SCr greater than or equal to (>=) 6.0 mg/dL (530 micromoles/Liter; micromol/L) for >= 4 weeks as determined by the local laboratory; regularly scheduled dialysis treatments over a period of 56 days; impairment of renal function to such a degree that the participant undergoes re-transplant. Day 1 was day of transplantation. ITT population defined as all participants randomized and transplanted.
Time Frame: Day 1 to Month 6 and Month 12 post transplantation
Population: Participants surviving with a functioning graft were 30, 24, 30 in belatacept/MMF, belatacept/sirolimus, tacrolimus/MMF arms, respectively. Participant who died had functioning graft at time of death.
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 33 | 26 | 30
participants
  Graft loss up to Month 6 post transplantation | 1 | 1 | 0
  Graft loss up to Month 12 post transplantation | 2 | 2 | 0
  Death up to Month 6 post transplantation | 1 | 0 | 0
  Death up to Month 12 post transplantation | 1 | 0 | 0

4. Secondary Outcome: Number of Participants With Composite of Death, Graft Loss and Acute Rejection up to Month 6 - Intent to Treat Population
Description: Participants with graft loss or death prior to Month 6 were considered having an event of AR, therefore, the incidence of AR was reported as a composite of AR, death, and graft loss.
Time Frame: Day 1 up to Month 6
Population: Intent to treat population included all randomized and transplanted participants.
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 33 | 26 | 30
participants | 6 | 2 | 1

5. Secondary Outcome: Number of Participants With Composite of Death, Graft Loss and Acute Rejection up to Month 12 - Intent to Treat Population
Description: Subjects with graft loss or death prior to Month 12 were considered having an event of AR, therefore, the incidence of AR was reported as a composite of AR, death, and graft loss.
Time Frame: Day 1 up to Month 12
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 33 | 26 | 30
participants | 7 | 3 | 1

6. Secondary Outcome: Number of Participants With Delayed Graft Function - Intent to Treat Population
Description: Delayed graft function (DGF) is defined as participant requiring dialysis within the first week (Day 1-8) post transplantation. Participants losing their graft less than 48 hours post transplant and receiving chronic dialysis were not considered as having DGF. Day 1 was day of transplantation. Intent to treat population defined as all participants randomized and transplanted
Time Frame: From Day 1 up to and including Day 8 post transplantation
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 33 | 26 | 30
participants | 6 | 4 | 2

7. Secondary Outcome: Number of Participants With New Onset Diabetes Mellitus From Baseline to Month 12 Post Transplantation - Intent to Treat Population
Description: Baseline defined as day before transplantation. A participant who did not have diabetes prior to randomization and received an antidiabetic medication for a duration of at least 30 days or a participant who meets the following criteria and did not have diabetes prior to randomization: Symptoms of diabetes plus casual plasma glucose (PG) concentration ≥ 200 mg/dL (11.1 mmol/L); or fasting plasma glucose ≥ 126 mg/dL (7.0 mmol/L); or 2-hour PG ≥ 200 mg/dL (11.1 mmol/L) during an oral glucose tolerance test and a confirmatory laboratory test based on measurements of venous PG must have been done on another day in the absence of unequivocal hyperglycemia accompanied by acute metabolic decompensation.
  Intent to treat population included all participants randomized and transplanted.
Time Frame: Baseline to Month 12
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 33 | 26 | 30
participants | 0 | 2 | 1

8. Secondary Outcome: Number of Participants Who Used Anti-hypertension Medications at Baseline and at 12 Months Post Transplantation - Intent to Treat Population
Description: Baseline was defined as day prior to transplantation. Number of anti-hypertension medications taken were categorized from 1 to 6 and greater than (>)6. Intent to treat population included all participants randomized and transplanted.
Time Frame: Baseline and Month 12
Population: ITT population, 33, 26, 30 for each arm, respectively, was used for each time point (baseline and Month 12). At baseline, 2 participants in each arm were not using at least one medication. 8, 6, and 10 participants in each arm respectively, were not using at least one medication at Month 12.
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 33 | 26 | 30
participants
  Total using at least 1 medication at baseline | 31 | 24 | 28
  Total using at least 1 medication at Month 12 | 25 | 20 | 20
  Participants using 1 medication at baseline | 10 | 9 | 5
  Participants using 1 medication at Month 12 | 11 | 5 | 4
  Participants using 2 medications at baseline | 5 | 5 | 8
  Participants using 2 medications at Month 12 | 6 | 8 | 13
  Participants using 3 medications at baseline | 8 | 5 | 8
  Participants using 3 medications at Month 12 | 6 | 5 | 0
  Participants using 4 medications at baseline | 3 | 2 | 3
  Participants using 4 medications at Month 12 | 1 | 2 | 3
  Participants using 5 medications at baseline | 3 | 1 | 2
  Participants using 5 medications at Month 12 | 0 | 0 | 0
  Participants using 6 medications at baseline | 2 | 2 | 1
  Participants using 6 medications at Month 12 | 1 | 0 | 0
  Participants using >6 medications at baseline | 0 | 0 | 1
  Participants using >6 medications at Month 12 | 0 | 0 | 0

9. Secondary Outcome: Mean Systolic, Diastolic and Arterial Blood Pressure at Baseline and Month 12 - Intent to Treat Population
Description: Systolic, diastolic and mean arterial blood pressures were measured in millimeters of mercury (mm Hg). Baseline was defined as value obtained before transplantation. Intent to treat population included all participants randomized and transplanted.
Time Frame: Baseline and 12 months post transplantation
Population: Number analyzed at baseline presented above. Number analyzed at Month 12: 28, 22, 29 in belatacept/MMF, belatacept/sirolimus, and tacrolimus/MMF treatment arms,respectively. Measurements obtained immediately after drug infusion were excluded from analysis.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 33 | 26 | 30
mm Hg
  Systolic blood pressure at baseline | 133.1 (26.43) | 126.9 (18.72) | 141.8 (23.79)
  Systolic blood pressure at Month 12 | 129.3 (19.24) | 131.0 (19.88) | 138.2 (19.50)
  Diastolic blood pressure at baseline | 78.6 (12.50) | 72.3 (11.27) | 75.3 (15.08)
  Diastolic blood pressure at Month 12 | 73.3 (11.96) | 75.1 (10.71) | 77.6 (10.51)
  Mean Arterial pressure at baseline | 96.8 (15.60) | 90.5 (12.84) | 97.5 (15.87)
  Mean Arterial pressure at Month 12 | 91.9 (12.80) | 93.7 (11.64) | 97.8 (10.90)

10. Secondary Outcome: Number of Participants Using Antihyperlipidemic Medications at Month 12 - Intent to Treat Population
Description: Participants using > = 1 antihyperlipidemic medication at Month 12.
Time Frame: Month 12
Population: Analysis based on all participants who were followed up at least 364 days.
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 31 | 26 | 26
participants | 11 | 10 | 9

11. Secondary Outcome: Mean Change From Baseline (BL) to Month 12 Post Transplantation in Lipid Values - Intent to Treat Population
Description: Baseline (BL) was value obtained day prior to transplantation. Lipid values measured in milligrams/deciliter (mg/dL) included: high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C), non-HDL cholesterol (non-HDL-C), total cholesterol (TC), triglycerides. Intent to treat population included all participants randomized and transplanted.
Time Frame: Baseline to Month 12
Population: 33, 26, 30 participants were included in the ITT population. Number of participants analyzed for HDL-C = 26, 22, 26; non-HDL-C = 26, 22, 26; LDL-C = 20, 14, 21; TC = 26, 22, 26; triglycerides = 20, 14, 21, in belatacept/MMF, belatacept/sirolimus, and tacrolimus/MMF arms, respectively.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 33 | 26 | 30
mg/dL
  HDL-C change from BL to Month 12 | 1.5 (12.70) | -3.7 (12.94) | -0.5 (12.24)
  Non-HDL-C change from BL to Month 12 | 16.0 (45.25) | 16.1 (45.15) | 20.5 (42.56)
  LDL-C change from BL to Month 12 | 23.9 (38.18) | 25.0 (37.17) | 34.0 (30.18)
  Total cholesterol change from BL to Month 12 | 17.5 (40.69) | 12.5 (49.03) | 20.0 (45.80)
  Triglycerides change from BL to Month 12 | -11.4 (63.31) | -1.1 (88.88) | -14.2 (94.83)

12. Secondary Outcome: Mean (Standard Deviation) in Calculated Glomerular Filtration Rate (GFR) mL/Min/1.73m^2 at Month 3, Month 6 and Month 12 Post Transplantation - Intent to Treat Population
Description: Blood urea nitrogen (BUN) in mg/dL; Albumin (Alb) in g/dL;Serum creatinine (SCr) in mg/dL; Age in years. Glomerular filtration rate (GFR) was calculated based upon serum creatinine (SCr) using the Modification of Diet in Renal Disease (MDRD) formula as suggested by Levey et al: MDRD GFR = 170 x [SCr/0.95]^(-0.999) x [Age]^(-0.176) x [0.762 if participant was female] x [1.180 if participant was black] x [BUN]^(-0.170) x [Alb]^(+0.318). Intent to Treat (ITT) population is defined as all participants randomized and transplanted.
Time Frame: Months 3, 6 and 12 post transplantation
Population: Month 12 n presented above. Calculated GFR, values >180 mL/min/1.73 m2 (beyond upper limit of biologic plausibility)were truncated at 180 mL/min/1.73 m^2. Based on median (SD) GFR of 83 (50).
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 29 | 24 | 29
mL/min/1.73m^2
  Month 3 post transplantation(n=29,24,27) | 57.8 (15.41) | 60.5 (26.69) | 51.2 (14.78)
  Month 6 post transplantation(n=29,24,25) | 57.5 (14.75) | 58.7 (28.36) | 51.7 (17.80)
  Month 12 post transplantation(n=27, 23, 29) | 63.6 (27.27) | 61.8 (30.66) | 54.0 (14.95)

13. Secondary Outcome: Number of Corticosteroid-free Participants at 6 and 12 Months Post Transplantation - Intent to Treat Population
Description: Participants were said to be corticosteroid-free at Month 6 if they were not receiving corticosteroids for greater than (>) 7 consecutive days during Days 141 through Days 196, and at Month 12 if not receiving corticosteroids for > 7 days during Days 337 through 392. Intent to treat population included all randomized and transplanted participants.
Time Frame: Day 1 through Month 12
Population: For 95% CI within each group, normal approximation was used if N greater than, equal to (>=)5. Otherwise, exact method was used. Numbers of participants analyzed at Month 6 in each arm were 33, 26, 30 and numbers of participants analyzed at Month 12 were 32, 26, 30, in belatacept/MMF, belatacept/sirolimus, and tacrolimus/MMF arms, respectively.
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 33 | 26 | 30
participants
  At 6 Months post transplantation | 27 [68.7 to 95.0] | 23 [76.2 to 100.0] | 28 [84.4 to 100.0]
  At 12 Months post transplantation | 24 [60.0 to 90.0] | 20 [60.7 to 93.1] | 28 [84.4 to 100.0]

14. Secondary Outcome: Number of Participants Who Were Corticosteroid-free at Months 6 and 12 and Number of Participants Who Were Both Calcineurin Inhibitor-free (CNI-free)and Corticosteroid-free at Months 6 and 12 Post Transplantation - Intent to Treat Population
Description: Participants were said to be CNI-free at Month 6 or 12 if they were not receiving a CNI during Day 141 to Day 196, or Day 337 to Day 392. Participants in the tacrolimus arm were not relevant to this analysis because tacrolimus is a calcinurin inhibitor. Participants were corticosteroid-free (CS-free) at Month 6 if they were not receiving corticosteroids for > 7 consecutive days during Days 141 through Days 196, and at Month 12 if not receiving corticosteroids for > 7 days during Days 337 through 392. Day 1 was day of transplantation. Intent to treat population included all randomized and transplanted participants.
Time Frame: Day 1 to Month 12 post transplantation
Population: Analysis on both CNI-free and CS-free participants based on all followed up at least 151 days for Month 6 or 347 days for Month 12. One participant in the tacrolimus arm was counted as CNI-free since he discontinued tacrolimus on Day 2 of transplant and no data were available regarding immunosuppressive therapy after discontinuation.
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 33 | 26 | 30
participants
  CS-free Month 6 (N=33, 26, 30) | 27 | 23 | 28
  CS-free Month 12 (N=32, 26, 30) | 24 | 20 | 28
  CNI-free + CS-free Month 6 (N=32, 26, 30) | 25 | 19 | 1
  CNI -free + CS-free Month 12 (N=32,26,30) | 24 | 18 | 1

15. Secondary Outcome: Number of Participants With Acute Rejection of Transplant up to End of Month 48 Post Transplantation - Intent to Treat Population in Long Term Extension
Description: as for outcome 2
Time Frame: End of Month 12 to end of Month 48 Post Transplantation
Population: All participants who completed the short term (ST) period, were eligible and accepted to enter the LTE by signing a new informed consent form.
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 27 | 19 | 27
participants | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Graft Loss or Death at Months 24, 36, 48 Post Transplantation - Intent to Treat Population in Long Term Extension
Description: as for outcome 3
Time Frame: End of Month 12 to end of Long Term Extension (Year 4)
Population: N=participants randomized and transplanted and in LTE.
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 27 | 19 | 27
participants
  Graft Loss or Death at Month 24 (N=27,19,27) | 0 | 1 | 0
  Graft Loss or Death at Month 36 (N=27,19,27) | 1 | 2 | 0
  Graft Loss or Death at Month 48 (N=27,19,27) | 1 | 2 | 0

17. Secondary Outcome: Mean (Standard Deviation) in Calculated Glomerular Filtration Rate (GFR) mL/Min/1.73m^2 at Months 24, 36 and 48 Post Transplantation - Intent to Treat Population in Long Term Extension
Description: GFR was calculated based upon serum creatinine (SCr) using the Modification of Diet in Renal Disease (MDRD) formula as suggested by Levey et al: MDRD GFR = 170 x [SCr/0.95]^(-0.999) x [Age]^(-0.176) x [0.762 if participant was female] x [1.180 if participant was black] x [BUN]^(-0.170) x [Alb]^(+0.318). Age in years, Alb = Albumin in g/dL; SCr = in mg/dL; BUN =Blood urea nitrogen in mg/dL. Intent to Treat population is defined as all participants randomized and transplanted.
Time Frame: Months 24, 36 and 48 post transplantation
Population: N=All participants who were randomized, transplanted, in the LTE and had data available at the specific time point.
Measure: Mean (Standard Deviation); unit: mL/Min/1.73m^2
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 27 | 18 | 27
mL/Min/1.73m^2
  Month 24 (N=27, 18, 27) | 60.6 (15.12) | 66.0 (23.75) | 52.2 (12.14)
  Month 36 (N=25, 16, 22) | 62.8 (14.05) | 69.9 (22.43) | 55.5 (15.38)
  Month 48 (N=18, 14, 15) | 59.6 (15.30) | 72.2 (25.21) | 55.7 (13.47)

18. Secondary Outcome: Number of Corticosteroid-free Participants at Months 24, 36, 48 Post Transplantation - Intent to Treat Population in Long Term Extension
Description: In the LTE, a participant was considered corticosteroid-free if they were not receiving corticosteroids for >7 consecutive days during Day 701 and Day 756, Day 1065 and Day 1120, as well as Day 1429 and Day 1484, respectively.
Time Frame: End of Month 12 to end of Long Term Extension (Year 4)
Population: N= All participants who completed the ST period, were eligible and accepted to enter the LTE by signing a new informed consent form, and had data available at the specific time point were analyzed.
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 27 | 18 | 27
participants
  Month 24 (N=27, 18, 27) | 22 | 15 | 25
  Month 36 (N=26, 16, 23) | 22 | 14 | 20
  Month 48 (N=19, 14, 16) | 16 | 12 | 16

19. Secondary Outcome: Number of Participants Who Were Both Calcineurin Inhibitor-free (CNI-free)and Corticosteroid-free at Months 24, 36, 48 Post Transplantation - Intent to Treat Population in Long Term Extension
Description: Participants were considered corticosteroid-free at Months 24, 36, and 48 if they were not receiving corticosteroids for >7 consecutive days during Day 701 and Day 756, Day 1065 and Day 1120, as well as Day 1429 and Day 1484, respectively. Participants were considered CNI-free at Months 24, 36, and 48 if they were not receiving CNI during Day 701 and Day 756, Day 1065 and Day 1120, as well as Day 1429 and Day 1484, respectively. Participants in the tacrolimus arm were not relevant to this analysis because tacrolimus is a calcinurin inhibitor.
Time Frame: Months 24, 36, 48
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 27 | 18 | 27
participants
  Month 24 (N=27, 18, 27) | 22 | 15 | 0
  Month 36 (N=26, 16, 23) | 22 | 14 | 0
  Month 48 (N=19, 14, 16) | 16 | 12 | 0

20. Secondary Outcome: Number of Participants Who Switched Between MMF and Sirolimus During Long Term Extension up to Study Completion
Description: Long Term extension was the period from the end of Month 12 to the end of Month 48 post transplantation and the completion of the study 31 July 2012. At any time in the study, participants who were unable to tolerate MMF in the Bela-MMF and Tac-MMF groups could discontinue (DC) MMF and switch to sirolimus and remain in the study and those in the Bela-Siro group who were unable to tolerate sirolimus could DC sirolimus and switch to MMF and remain in the study. Study completion=data base (DB) lock.
Time Frame: End of Month 12 to end of Study (Month 48)
Population: N= All participants who completed the ST period, were eligible and accepted to enter the LTE by signing a new informed consent form
Measure: Number; unit: participants
Arm/Group | Belatacept, Mycophenolate Mofetil (MMF) | Belatacept, Sirolimus | Tacrolimus, MMF
Number analyzed (Participants) | 27 | 19 | 27
participants
  By Month 24 Switched between MMF and Sirolimus | 0 [0 to 0] | 1 [0.1 to 26.0] | 0 [0 to 0]
  By Month 36 Switched between MMF and Sirolimus | 0 [0 to 0] | 2 [1.3 to 33.1] | 0 [0 to 0]
  By Month 48 Switched between MMF and Sirolimus | 0 [0 to 0] | 3 [3.4 to 39.6] | 0 [0 to 0]
  Up to DB Lock Switched between MMF and Sirolimus | 0 [0 to 0] | 3 [3.4 to 39.6] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: From Day 1 to end of 48 Months post transplantation and study closure
Description: Total population of randomized participants in both short term period and long term extension.
Arm/Group | Belatacept - MMF | Belatacept - SIRO | Tacrolimus - MMF
Serious Adverse Events (participants affected / at risk) | 25/33 | 19/26 | 22/30
Other Adverse Events (participants affected / at risk) | 33/33 | 26/26 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept - MMF (N=33) | Belatacept - SIRO (N=26) | Tacrolimus - MMF (N=30)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Cytomegalovirus viraemia (Infections and infestations) | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 0 | 1 | 2
Graft loss (Injury, poisoning and procedural complications) | 1 | 1 | 0
Herpes zoster ophthalmic (Infections and infestations) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Renal artery thrombosis (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 1
Splenic abscess (Infections and infestations) | 0 | 0 | 1
Urinary fistula (Renal and urinary disorders) | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 2 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Ureteric dilatation (Renal and urinary disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 1
Chills (General disorders) | 0 | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0
Hyperpyrexia (General disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 1
Encephalitis herpes (Infections and infestations) | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Fungaemia (Infections and infestations) | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 2 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Secondary amyloidosis (Immune system disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 2
Urosepsis (Infections and infestations) | 0 | 0 | 2
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 4
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 2
Device malfunction (General disorders) | 0 | 1 | 0
Encephalitis fungal (Infections and infestations) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Renal vein thrombosis (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastrointestinal amyloidosis (Gastrointestinal disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 2 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Lymphocele (Vascular disorders) | 1 | 1 | 0
Meningitis cryptococcal (Infections and infestations) | 1 | 0 | 0
Mitral valve stenosis (Cardiac disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept - MMF (N=33) | Belatacept - SIRO (N=26) | Tacrolimus - MMF (N=30)
Abdominal pain lower (Gastrointestinal disorders) | 6 | 2 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 4 | 9 | 0
Blood glucose increased (Investigations) | 0 | 0 | 2
Blood iron decreased (Investigations) | 1 | 2 | 0
Blood urine present (Investigations) | 2 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 16 | 11 | 12
Diarrhoea (Gastrointestinal disorders) | 13 | 17 | 21
Dizziness (Nervous system disorders) | 5 | 4 | 6
Electrolyte imbalance (Metabolism and nutrition disorders) | 3 | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 2
Face oedema (General disorders) | 2 | 2 | 3
Fluid retention (Metabolism and nutrition disorders) | 2 | 2 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 3 | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 0 | 1 | 4
Haematochezia (Gastrointestinal disorders) | 4 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 4 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Insomnia (Psychiatric disorders) | 7 | 5 | 7
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 4 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 4 | 4 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Renal tubular necrosis (Renal and urinary disorders) | 3 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 1
Urine output decreased (Investigations) | 2 | 2 | 3
Vomiting (Gastrointestinal disorders) | 11 | 5 | 8
Weight decreased (Investigations) | 6 | 6 | 4
Amnesia (Nervous system disorders) | 2 | 1 | 3
Asthenia (General disorders) | 10 | 8 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 8 | 4
Blood pressure increased (Investigations) | 3 | 0 | 6
Conjunctivitis (Eye disorders) | 2 | 1 | 0
Disturbance in attention (Nervous system disorders) | 2 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Headache (Nervous system disorders) | 7 | 9 | 9
Hyperparathyroidism (Endocrine disorders) | 3 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 12 | 6 | 5
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0 | 3
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3 | 4
Pyrexia (General disorders) | 16 | 17 | 15
Renal impairment (Renal and urinary disorders) | 0 | 2 | 4
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Sinus headache (Nervous system disorders) | 3 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Tooth infection (Infections and infestations) | 3 | 1 | 1
Toothache (Gastrointestinal disorders) | 2 | 3 | 1
Ureteric dilatation (Renal and urinary disorders) | 0 | 0 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
White blood cell count decreased (Investigations) | 2 | 2 | 3
White blood cell count increased (Investigations) | 2 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 7
Blood creatinine increased (Investigations) | 6 | 3 | 7
Chills (General disorders) | 6 | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 4
Dyslipidaemia (Metabolism and nutrition disorders) | 7 | 3 | 2
Dysuria (Renal and urinary disorders) | 4 | 1 | 4
Hot flush (Vascular disorders) | 2 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 5 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 4 | 6
Hyperparathyroidism tertiary (Endocrine disorders) | 1 | 0 | 2
Hypertension (Vascular disorders) | 11 | 9 | 13
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 2 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Laceration (Injury, poisoning and procedural complications) | 1 | 2 | 3
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Localised infection (Infections and infestations) | 3 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 3 | 8 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Nasopharyngitis (Infections and infestations) | 8 | 7 | 4
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Pain (General disorders) | 1 | 4 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 7 | 5
Procedural pain (Injury, poisoning and procedural complications) | 19 | 11 | 13
Renal disorder (Renal and urinary disorders) | 1 | 0 | 2
Scrotal oedema (Reproductive system and breast disorders) | 2 | 2 | 1
Sinusitis (Infections and infestations) | 6 | 4 | 4
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Bronchitis (Infections and infestations) | 4 | 1 | 0
Depression (Psychiatric disorders) | 3 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Fungal infection (Infections and infestations) | 0 | 0 | 2
Hypotension (Vascular disorders) | 7 | 4 | 4
Influenza (Infections and infestations) | 3 | 2 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Lethargy (Nervous system disorders) | 2 | 0 | 2
Micturition urgency (Renal and urinary disorders) | 2 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Oral candidiasis (Infections and infestations) | 2 | 3 | 0
Oral herpes (Infections and infestations) | 4 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 1
Pneumonia (Infections and infestations) | 2 | 2 | 1
Prostatic specific antigen increased (Investigations) | 1 | 0 | 2
Proteinuria (Renal and urinary disorders) | 6 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 2
Vision blurred (Eye disorders) | 2 | 1 | 5
Wound (Injury, poisoning and procedural complications) | 1 | 2 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 4
Anaemia (Blood and lymphatic system disorders) | 20 | 18 | 14
Anxiety (Psychiatric disorders) | 4 | 6 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Bladder spasm (Renal and urinary disorders) | 4 | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 6
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 4 | 3 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Incision site haemorrhage (Injury, poisoning and procedural complications) | 2 | 0 | 3
Malaise (General disorders) | 2 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Odynophagia (Gastrointestinal disorders) | 1 | 3 | 0
Oedema peripheral (General disorders) | 14 | 15 | 10
Parathyroid gland enlargement (Endocrine disorders) | 0 | 0 | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Renal bruit (Investigations) | 1 | 0 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sleep disorder (Psychiatric disorders) | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 14 | 8 | 10
Abdominal tenderness (Gastrointestinal disorders) | 1 | 2 | 4
Bloody discharge (Vascular disorders) | 1 | 1 | 2
Breath sounds abnormal (Investigations) | 5 | 2 | 5
Cataract (Eye disorders) | 0 | 2 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 2
Fatigue (General disorders) | 7 | 8 | 9
Furuncle (Infections and infestations) | 1 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 6 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 2
Oedema (General disorders) | 5 | 3 | 3
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Tachycardia (Cardiac disorders) | 5 | 5 | 2
Urethral stenosis (Renal and urinary disorders) | 1 | 2 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 2
Weight increased (Investigations) | 6 | 4 | 7
Abdominal distension (Gastrointestinal disorders) | 2 | 4 | 4
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
BK virus infection (Infections and infestations) | 2 | 1 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 5 | 4 | 5
Dry eye (Eye disorders) | 0 | 1 | 2
Ear infection (Infections and infestations) | 1 | 2 | 3
Generalised oedema (General disorders) | 3 | 4 | 5
Haemoglobin decreased (Investigations) | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 6 | 2 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 8 | 4
Incision site erythema (Injury, poisoning and procedural complications) | 2 | 2 | 4
Incision site pain (Injury, poisoning and procedural complications) | 4 | 5 | 7
Leukopenia (Blood and lymphatic system disorders) | 18 | 12 | 15
Lymphopenia (Blood and lymphatic system disorders) | 3 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 2 | 1
Paraesthesia (Nervous system disorders) | 4 | 3 | 4
Polycythaemia (Blood and lymphatic system disorders) | 2 | 0 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 2 | 3
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 9 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Cellulitis (Infections and infestations) | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 5
Cytomegalovirus infection (Infections and infestations) | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 5 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Gastroenteritis (Infections and infestations) | 2 | 2 | 0
Haematuria (Renal and urinary disorders) | 9 | 11 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 4 | 4
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1
Memory impairment (Nervous system disorders) | 2 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 14 | 7 | 12
Neuropathy peripheral (Nervous system disorders) | 2 | 1 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 5 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 2
Seasonal allergy (Immune system disorders) | 3 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 9
Urinary retention (Renal and urinary disorders) | 2 | 1 | 3

LIMITATIONS AND CAVEATS:
Main limitations of this study include: small size (small number of participants in each treatment arm), the open-label nature of the trial, its exploratory nature, and the high rate of switches from sirolimus to MMF in one of the belatacept groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.